CLINICAL TRIAL: NCT07395700
Title: Psychometric Validation of the Behavioral Activation for Depression Scale (BADS) in a Clinical Sample of Individuals With Substance Use Disorders
Brief Title: Validation of the Behavioral Activation for Depression Scale in Individuals With Substance Use Disorders
Acronym: BADS-SUD
Status: Completed | Type: Observational
Sponsor: Lauro Gutiérrez Castro (Other)
Responsible Party: Sponsor-Investigator, Lauro Gutiérrez Castro, Principal Invetigator, Under The Tree Therapeutic Community
Organization: Under The Tree Therapeutic Community (Other)
Other Study IDs: BADS-SUD-VALID-01
Record Dates: First submitted 2026-01-07; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Substance Use Disorders; Mental Health Disorders; Substance-related Disorders; Depression Scale Score; Validation Study
Keywords: Behavioral Activation; Psychometric Validation; Substance Use Disorders; Addiction; External Validity; Incremental Validity; Clinical Assessment; Behavioral Functioning; Depression; Functional Impairment
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals With Substance Use Disorders: Single clinical group composed of adults receiving treatment for substance use disorders who completed the Behavioral Activation for Depression Scale (BADS) and additional self-report measures as part of a cross-sectional observational study.

SUMMARY:
This observational study evaluates the psychometric properties of the Behavioral Activation for Depression Scale (BADS) in individuals with substance use disorders. The study examines the scale's internal structure, reliability, and validity using data from 289 participants who completed the BADS. External and incremental validity analyses were conducted in a subsample of 127 participants for whom additional clinical measures were available, including assessments of symptom severity, anxiety, impulsivity, and anger expression. This approach reflects the availability of complete data for each analytic component and allows for a comprehensive evaluation of the BADS in a clinical population.

DETAILED DESCRIPTION:
This study employs a cross-sectional observational design to evaluate the psychometric performance of the Behavioral Activation for Depression Scale (BADS) in individuals with substance use disorders. The validation process consisted of two complementary analytic components based on data availability.

First, analyses of internal structure, reliability, and item-level performance were conducted using data from 289 participants who completed the BADS. These analyses included advanced psychometric methods to evaluate the dimensional structure and measurement properties of the scale.

Second, external and incremental validity analyses were conducted in a subsample of 127 participants for whom complete data were available on additional validated self-report measures assessing clinically relevant constructs, including symptom severity, anxiety, impulsivity, and anger expression. This subsample approach reflects the naturalistic data collection process in clinical settings and allowed for the examination of the BADS' relationships with external criteria without imputing missing data.

Together, these analyses provide a comprehensive evaluation of the BADS, integrating evidence from internal psychometric validation and external criterion-related validity in a clinical population with substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Currently receiving treatment or undergoing clinical evaluation for substance use disorders in a therapeutic or clinical setting.
* Ability to read and understand Spanish.
* Ability to provide informed consent.
* Completion of the Behavioral Activation for Depression Scale and at least one additional study questionnaire.

Exclusion Criteria:

* Severe cognitive impairment or acute psychiatric symptoms that prevent accurate self-reporting.
* Incomplete or missing data on key study measures.
* Current intoxication or acute withdrawal symptoms at the time of assessment that interfere with completing questionnaires.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults receiving residential treatment for substance use disorders in a therapeutic community setting. Participants represent a clinically relevant population characterized by difficulties in mood regulation, behavioral activation, emotional dysregulation, and related psychological symptoms commonly associated with substance use disorders.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Psychometric Validity of the Behavioral Activation for Depression Scale (BADS) | Baseline, pre-intervention (single cross-sectional assessment at study enrollment)
  Psychometric properties of the Behavioral Activation for Depression Scale (BADS), including internal structure (confirmatory factor analysis), internal consistency reliability (Cronbach's alpha / omega), and construct validity (convergent and discriminant validity), assessed using self-report data collected at a single time point in individuals with substance use disorders. Subscale scores will also be examined, with higher scores reflecting greater expression of the respective behavioral domains.

SECONDARY OUTCOMES:
Convergent and Discriminant Validity of the Behavioral Activation for Depression Scale With the Borderline Symptom List-23 | Baseline, pre-intervention (single cross-sectional assessment conducted at study enrollment)
  Convergent and discriminant validity of the Behavioral Activation for Depression Scale will be examined through its association with scores on the Borderline Symptom List-23, a self-report measure of borderline symptom severity and behavioral dysregulation. The Borderline Symptom List-23 provides a mean total score ranging from 0 to 4, with higher scores indicating greater severity of borderline symptomatology. Associations will be analyzed using continuous scores to evaluate the extent to which behavioral activation and avoidance patterns measured by the Behavioral Activation for Depression Scale relate to clinical severity and emotional dysregulation in individuals with substance use disorders. The Borderline Symptom List-23 is a 23-item self-report scale scored on a 5-point Likert-type format (0 to 4), producing a mean total score ranging from 0 to 4. Higher scores indicate greater severity of borderline symptomatology and emotional dysregulation.
Convergent Validity of the Behavioral Activation for Depression Scale With the Environmental Reward Observation Scale | Baseline, pre-intervention (single cross-sectional assessment at study enrollment)
  Convergent validity of the Behavioral Activation for Depression Scale will be evaluated through its association with the Environmental Reward Observation Scale, a self-report measure assessing perceived availability and frequency of environmental positive reinforcement. The Environmental Reward Observation Scale consists of 10 items scored on a Likert-type scale, with higher total scores reflecting greater perceived environmental reinforcement. Correlations between Behavioral Activation for Depression Scale scores and Environmental Reward Observation Scale scores will be analyzed as continuous variables to examine the theoretical correspondence between behavioral activation processes and perceived environmental reinforcement in a residential substance use treatment context. The Environmental Reward Observation Scale consists of 10 items scored on a 4-point Likert-type scale, yielding total scores ranging from 10 to 40, with higher scores indicating greater perceived availability of en

CONTACTS AND LOCATIONS:
Overall Officials: Lauro Gutiérrez Castro, Principal Investigator — Under The Tree Therapeutic Community
Locations (1):
- Comunidad Terapéutica Under The Tree, Ajijic, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No